CLINICAL TRIAL: NCT06256913
Title: Phénogroupage basé Sur l'Apprentissage Automatique Dans la Cardiomyopathie Hypertrophique Pour Identifier Les Facteurs prédictifs de la Fibrose Myocardique et Les événements Cardiovasculaires
Brief Title: Machine Learning Approach Based on Echocardiographic Data to Improve Prediction of Cardiovascular Events in Hypertrophic Cardiomyopathy
Acronym: 2022PI172
Status: Recruiting | Type: Observational
Sponsor: Pr. Nicolas GIRERD (Other)
Responsible Party: Sponsor-Investigator, Pr. Nicolas GIRERD, Clinical Professor, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Other Study IDs: 2022PI172
Record Dates: First submitted 2024-01-16; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with sarcomeric hypertrophic cardiomyopathy and cardiovascular events: Patients with confirmed sarcomeric hypertrophic cardiomyopathy who experienced cardiovascular events.
- Patients with sarcomeric hypertrophic cardiomyopathy free of cardiovascular events: Patients with confirmed sarcomeric hypertrophic cardiomyopathy free of cardiovascular events.

SUMMARY:
Hypertrophic cardiomyopathy is a pathology with a highly variable course, ranging from patients who are asymptomatic throughout their lives to those who experience sudden death and/or terminal heart failure.

The main objective is to develop and validate an algorithm (constructed through supervised learning) using cardiac imaging data to predict the risk of cardiovascular events in sarcomeric hypertrophic cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Patients with confirmed sarcomeric hypertrophic cardiomyopathy

Exclusion Criteria:

* Echocardiographic data not allowing deep analysis (technical default, bad echogenicity of the patient)
* Other causes of left ventricular hypertrophy that may hamper the diagnosis (p.e. aortic or sub-aortic stenosis, severe renal insufficiency, hypertension).
* History of ischemic heart disease or associated myocarditis
* Opposition of the patient to the use of his/her data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Confirmed sarcomeric hypertrophic cardiomyopathy population
Sampling Method: Non-Probability Sample
Enrollment: 870 (Estimated)
Dates: Start 2023-05-06 (Actual); Primary Completion 2024-05-06 (Estimated); Study Completion 2024-05-06 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular mortality (composite) | From date of start of follow-up until death or loss to follow-up (up to 12 years of FU)
  Rates of cardiovascular mortality, hospitalisation for cardiovascular event, worsening of NYHA stage, onset of ventricular arrhythmia, onset of supra ventricular arrhythmia, onset of peripheral embolisms (stroke, TIA or acute limb ischemia) (With outcome 2,3,4,5,6)
Hospitalisation for cardiovascular event (composite) | From date of start of follow-up until death or loss to follow-up (up to 12 years of FU)
  Rates of cardiovascular mortality, hospitalization for cardiovascular event, worsening of NYHA stage, onset of ventricular arrhythmia, onset of supra ventricular arrhythmia, onset of peripheral embolisms (stroke, TIA or acute limb ischemia) (With outcome 1,3,4,5,6)
Worsening of NYHA stage (composite) | From date of start of follow-up until death or loss to follow-up (up to 12 years of FU)
  Proportion of cardiovascular mortality, hospitalisation for cardiovascular event, worsening of NYHA stage, onset of ventricular arrhythmia, onset of supra ventricular arrhythmia, onset of peripheral embolisms (stroke, TIA or acute limb ischemia) (With outcome 1,2,4,5,6)
Onset of ventricular arrhythmia (composite) | From date of start of follow-up until death or loss to follow-up (up to 12 years of FU)
  Proportion of cardiovascular mortality, hospitalisation for cardiovascular event, worsening of NYHA stage, onset of ventricular arrhythmia, onset of supra ventricular arrhythmia, onset of peripheral embolisms (stroke, TIA or acute limb ischemia) (With outcome 1, 2,3, 5,6)
Onset of supra ventricular arrhythmia (composite) | From date of start of follow-up until death or loss to follow-up (up to 12 years of FU)
  Proportion of cardiovascular mortality, hospitalisation for cardiovascular event, worsening of NYHA stage, onset of ventricular arrhythmia, onset of supra ventricular arrhythmia, onset of peripheral embolisms (stroke, TIA or acute limb ischemia) (With outcome 1, 2,3,4,6)
Onset of peripheral embolisms (stroke, TIA or acute limb ischemia) (composite) | From date of start of follow-up until death or loss to follow-up (up to 12 years of FU)
  Proportion of cardiovascular mortality, hospitalisation for cardiovascular event, worsening of NYHA stage, onset of ventricular arrhythmia, onset of supra ventricular arrhythmia, onset of peripheral embolisms (stroke, TIA or acute limb ischemia) (With outcome 1,2,3,4,5)

SECONDARY OUTCOMES:
Onset of tachycardia and or atrial fibrillation | From date of start of follow-up until death or loss to follow-up (up to 12 years of FU)
  Tachycardia and/or ventricular fibrillation during follow-up as well as sudden death, recovered or not recovered. (With outcome 8)
Sudden death, recovered or not recovered | From date of start of follow-up until death or loss to follow-up (up to 12 years of FU)
  Tachycardia and/or ventricular fibrillation during follow-up as well as sudden death, recovered or not recovered. (With outcome 7)
Cardiac decompensation requiring IV diuretics intake | From date of start of follow-up until death or loss to follow-up (up to 12 years of FU)
  Composite endpoint: cardiac decompensation requiring IV diuretics intake (managed in conventional hospitalization, day hospitalization or in-home) and the occurrence of atrial fibrillation, atrial tachycardia or atrial flutter. (With outcome 10)
Occurrence of atrial fibrillation, atrial tachycardia or atrial flutter | From date of start of follow-up until death or loss to follow-up (up to 12 years of FU)
  Composite endpoint: cardiac decompensation requiring IV diuretics intake (managed in conventional hospitalization, day hospitalization or in-home) and the occurrence of atrial fibrillation, atrial tachycardia or atrial flutter. (With outcome 9)
Cardiac remodelling | From date of start of follow-up until death or loss to follow-up (up to 12 years of FU)
  Evaluated by measurement of left ventricular mass as well as the appearance of late enhancement on MRI.
Cardiac remodelling | From date of start of follow-up until death or loss to follow-up (up to 12 years of FU)
  Evaluated by measurement of volume as well as the appearance of late enhancement on MRI.
Cardiac remodelling | From date of start of follow-up until death or loss to follow-up (up to 12 years of FU)
  Evaluated by measurement of function as well as the appearance of late enhancement on MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Girerd, MD, Study Chair — CHRU de Nancy
Locations (2):
- France (2):
  - CHU de Boredeaux Hôpital Cardiologique du Haut-Lévêque, Bordeaux
  - CHRU de Nancy, Nancy